CLINICAL TRIAL: NCT03168880
Title: A Randomized Controlled Trial of Neoadjuvant Weekly Paclitaxel Versus Weekly Paclitaxel Plus Weekly Carboplatin In Women With Large Operable or Locally Advanced, Triple Negative Breast Cancer
Acronym: TNBC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Rajendra A. Badwe, Director, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRI/2012/07/002802
Record Dates: First submitted 2017-05-20; First posted 2017-05-30 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — CP protocol

STUDY DESIGN:
Intervention Model Description: The study will test platinum based chemotherapy against the standard taxane based chemotherapy in the neo adjuvant setting as below:
  Arm A: Paclitaxel (weekly *8) + AE/EC 3 weekly *4 followed by Surgery + RT Arm B: Paclitaxel+ Carboplatin (weekly *8) + AE/EC 3 weekly *4 followed by Surgery+ RT
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): weekly Paclitaxel chemotherapy at the dose of 100 mg/m2/week for 8 weeks as a 1-hour infusion and AC/EC (60/600 or 90/600) / 3 weekly.
  Interventions: Drug: Paclitaxel only
- B (Experimental): weekly Paclitaxel at 100mg /m2/week + weekly Carboplatin AUC-2 as an infusion over 60 minutes and AC/EC (60/600 or 90/600)/ 3 weekly.
  Interventions: Drug: Paclitaxel + Carboplatin

INTERVENTIONS:
Drug: Paclitaxel + Carboplatin — Platinum based chemotherapy against the standard taxane based chemotherapy in the neo- adjuvant setting
  Arms: B
Drug: Paclitaxel only
  Arms: A

SUMMARY:
Triple-negative breast cancer is a subtype of breast cancer that is clinically negative for expression of estrogen and progesterone receptors (ER/PR) and HER2 protein. It is characterized by its unique molecular profile, aggressive behavior, distinct patterns of metastasis, and lack of targeted therapies. Although not synonymous, the majority of triple-negative breast cancers carry the "basal-like" molecular profile on gene expression arrays.

Although sensitive to chemotherapy, early relapse is common and these cancers show a predilection for visceral metastasis, including brain metastasis. Targeted agents, including epidermal growth factor receptor (EGFR), vascular endothelial growth factor (VEGF), and poly (ADP-ribose) polymerase (PARP) inhibitors, are currently in clinical trials and hold promise in the treatment of this aggressive disease.

Multiple independent data sets have revealed that the triple negative type of breast cancer carries a poor prognosis. It is unclear whether the poor prognosis of triple negative breast cancer is due to poor therapy options or inherent aggressiveness. Given their triple negative receptor status, these tumors are not amenable to conventional targeted therapies for breast cancer, such as endocrine therapy or trastuzumab, leaving only chemotherapy in the therapeutic armamentarium.

Patients on metformin showed a 30-40% protection against all forms of cancer. Recent pilot studies carried out using population registries raise the possibility that metformin may reduce cancer risk and/or improve cancer prognosis. One showed an unexpectedly lower risk of a cancer diagnosis among diabetics using metformin compared with a control group of diabetics using other treatments ; another showed lower cancer-specific mortality among subjects with diabetes using metformin compared with diabetics on other treatments. Metformin is a biguanide known to be an insulin sensitizing agent which promotes reduced circulating insulin and glucose levels in hyper-glycaemic and hyper-insulinaemic patients. Metformin activates the AMP dependent kinase, attenuates insulin and IGF-1 stimulated proliferation in breast cancer cells and a general decrease in protein synthesis in vitro. Western blot analysis indicated that metformin stimulates AMPK phosphorylation in a dose-dependent manner. AMPK activation is associated with decreased phosphorylation of mTOR and S6 kinase. While metformin reduces breast carcinoma cell proliferation both in vitro and in vivo, the activation of AMPK leads to significant VEGF production, angiogenesis and tumor progression. This must be taken into consideration when it is applied in as a therapeutic regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. All patients with baseline clinical staging T4, N0-3, M0 or T1-4, N2-3, M0 and T3, N1, M0 with triple negative hormone status.
3. Patients with adequate baseline marrow function defined as ANC > 1500/mm3 and Platelet count > 1, 00,000/mm3.
4. Patients with acceptable liver function tests (normal bilirubin and AST/ALT < 2 times the upper limit of normal) and normal renal function tests at baseline
5. Patients willing to provide informed consent
6. Patients fit for chemotherapy

Exclusion Criteria:

1. Prior excision biopsy
2. Metastatic breast cancer
3. Women with inflammatory breast cancer
4. Poor cardiac function at baseline with LVEF <40%
5. Patients with a prior history of a malignancy
6. Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2010-04; Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
DFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Disease free survival
OS | From date of randomization to the date of death or up to date of last follow-up for alive patients whichever came first, assessed up to 60 months
  Overall survival

OTHER OUTCOMES:
Response rate | 9-12 months from Randomization
  Clinical response evaluation during and at the end of Neo-adjuvant Chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Tata memorial Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided